CLINICAL TRIAL: NCT06348966
Title: Predictors of Hospital Readmission for Chronic Obstructive Pulmonary Disease Patients,A Prospective Cohort Study
Brief Title: Predictors of Hospital Readmission for Chronic Obstructive Pulmonary Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rougina Girgis Kamel Boles, resident doctor, Assiut University
Other Study IDs: predictors of readmission
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Hospital Radmission for COPD Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to determine the risk factors for hospital readmission within 6 months in COPD patients

DETAILED DESCRIPTION:
This study is aimed to determine the risk factors for hospital readmission within 6 months in COPD patients and develop early warning model

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients of both genders diagnosed by (GOLD) Guidelines (2024 Revision).
* Cooprative patients who accept to participate in the current study .

Exclusion Criteria:

* patients with cognitive impairment ,and unable to answer needed questions.
* patients with other lung diseases such as active pulmonary tuberculosis ,asthma ,bronchiactesis,and pulmonary embolism .
* patients with incomplete clinical data .
* Refused to participate in the current study .

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: this study is a prospective hospital-based cohort study
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
assessment of potential predictors of readmission among COPD patients | 6 months
  using CCI (charlson comorbidity index)

SECONDARY OUTCOMES:
development of early warning model for hospital readmission in COPD patients | within 6 months
  using CCI (charlson comorbidity index)

REFERENCES:
- [Background] Alqahtani JS, Aldabayan YS, Aldhahir AM, Al Rajeh AM, Mandal S, Hurst JR. Predictors of 30- and 90-Day COPD Exacerbation Readmission: A Prospective Cohort Study. Int J Chron Obstruct Pulmon Dis. 2021 Oct 7;16:2769-2781. doi: 10.2147/COPD.S328030. eCollection 2021. PMID 34675502
- [Background] Anbesse ZK, Mega TA, Tesfaye BT, Negera GZ. Early readmission and its predictors among patients treated for acute exacerbations of chronic obstructive respiratory disease in Ethiopia: A prospective cohort study. PLoS One. 2020 Oct 6;15(10):e0239665. doi: 10.1371/journal.pone.0239665. eCollection 2020. PMID 33022006